CLINICAL TRIAL: NCT06632899
Title: Effects of "Comprehensive Health Promotion and Healthy Lifestyle Development" in Community-dwelling Elderly.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 202400825B0
Record Dates: First submitted 2024-10-08; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-05

CONDITIONS: Community Centers
Keywords: Aged, community living elderly, active aging, multidomain interventions, health promotion, healthy lifestyle development.
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: combined physical and cognitive training and 1 hour of risk factor prevention and healthy lifestyle development
- control group (No Intervention)

INTERVENTIONS:
Behavioral: combined physical and cognitive training and 1 hour of risk factor prevention and healthy lifestyle development — Dosage: a 2-hour session once a week for 12 weeks. Each multidomain intervention session includes 1 hour of combined physical (balance, strength and aerobic exercises) and cognitive (attention, memory, calculation, visual-spatial ability, processing speed and executive function) training and 1 hour of risk factor prevention (nutrition, chronic disease management, oral health, fall prevention and transportation safety, psychosocial factors and sleep) and healthy lifestyle development (Discussion and sharing on topics such as self-health management, goal setting, and the "health journal.")
  Arms: intervention group

SUMMARY:
The World Health Organization (WHO) defines "Active Aging" as continued engagement in social, economic, cultural, spiritual, and civic activities, emphasizing the importance of participation for older adults. Personal health behaviors and habits influence both longevity and health status in later life, with healthy lifestyle development optimizing aging and enhancing well-being and quality of life.

WHO's Integrated Care for Older People (ICOPE) highlights six key indicators of physical and mental function-mobility, cognition, nutrition, vision, hearing, and depression-as critical to promoting active aging. These factors are also used to evaluate aging outcomes. Multidomain interventions are employed to address cognitive decline and dementia.

While research supports the benefits of multidomain interventions for cognitive improvement in older adults, consistent findings are lacking. Most interventions focus on exercise and cognitive training, with limited attention to other aging risk factors. Broader, more diverse interventions that actively involve older adults are needed to confirm the effects of these factors on cognitive function.

This study aims to evaluate the effects of multidomain interventions-covering exercise, cognitive training, nutrition, chronic disease management, vision and hearing care, fall prevention, psychosocial factors, and sleep-on mobility, cognition, daily functioning, and social participation in community-dwelling older adults

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old
2. Mini-Mental State Examination (MMSE) score > 20 (Folstein et al., 1975), able to follow instructions and participate in activities
3. With self-reported or caregiver-reported memory or cognitive-related problems
4. No diagnosis of any type of dementia

Exclusion Criteria:

1. Unstable medical condition that would prevent safe participation in exercise training (e.g., myocardial infarction, heart failure, recent cardiac surgery, severe asthma, concomitant neurological disorders, or joint deformities)
2. Participation in other studies
3. Inability to provide informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change scores of Montreal Cognitive Assessment (MoCA) | baseline, after the intervention 12 weeks
  The MoCA is used to assess general cognitive functions. It examines several cognitive domains with a total score of 30 and higher values indicate better cognitive functions. The MoCA has been shown to be a valid and promising tool to evaluate the global cognitive function in patients with stroke. The psychometric properties of MoCA are good to excellent for patients with cerebrovascular diseases.
Change scores of Timed up and go (TUG) | baseline, after the intervention 12 weeks
  The TUG assesses the dynamic balance ability and functional mobility. The participants will be required to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time to complete the TUG test has been shown to be a good indicator to detect potential fallers in frail elderly. The test-retest reliability of TUG on individuals with cognitive impairment is excellent.
Change scores of Grip strength (GS) | baseline, after the intervention 12 weeks
  Grip strength, a measure of body function, has been suggested as a biomarker of aging. The hand dynamometer is used to assess the upper limb strength of the participants. During the test, the participant's hand grips the handle with the second knuckle forming a right angle. The participant's elbow should be at a 90-degree angle, with their eyes looking straight ahead. The participant should squeeze the dynamometer tightly, ensuring it does not touch their body. GS assessment is a reliable and valid procedure among healthy participants as well as across various clinical populations.
Change scores of Outcome Measure of Health-Promotion Program for Community-Dwelling Elderly | baseline, after the intervention 12 weeks
  Outcome Measure of Health-Promotion Program for Community-Dwelling Elderly covers five dimensions: cognition, muscle strength, functional ability, nutrition and oral health, and psychosocial aspects. Each dimension consists of four questions, totaling 20 questions. This evaluation is designed to assess multidomain intervention and is suitable for elderly individuals with varying levels of ability, including healthy, frail, those with mild cognitive impairment, or mild to moderate disability/dementia. After conversion, the total score of this scale ranges from 0 to 100. A higher post-test score compared to the pre-test score indicates greater effectiveness in implementing the health promotion program. The 20-item health-promotion program outcome measure is concise and has good reliability/ validity.
Change scores of the Acting Aging Scale | baseline, after the intervention 12 weeks
  The Active Aging scale is administered through a questionnaire, utilizing a six-point Likert scale. The scale covers three dimensions: 1) "Health Promotion." 2) "Social Participation." 3) "Life Safety." Based on the participants' responses, six options ranging from "strongly disagree" to "strongly agree" are provided, with scores assigned from 1 to 6. A higher score indicates a higher level of active aging among the participants. the re-check validity of the measurement model was good, indicating that the scale could be applied to the senior population.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memotial Hospital, Taoyuan District, 龜山區, Taiwan

IPD SHARING:
Plan to Share IPD: No